CLINICAL TRIAL: NCT04646486
Title: Video Debriefing at the Delivery Ward - Empowering Obstetric Teams to High Performance
Brief Title: Video Debriefing at the Delivery Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Horsens Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEAMOBS Intervention
Record Dates: First submitted 2020-11-12; First posted 2020-11-30 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-09

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Data - videos of team performance - will be included as follows:
  Year 1) Baseline. Video inclusion, before introducing real-life video debriefings of team performance (n=200).
  Year 2) During the start-up of the debriefings (n=20) which will be evaluated in a feasibility study.
  Year 2-3) Intervention. After real-life video debriefings have been introduced as standard procedure (n=200).
Masking Description: Videos from baseline period and intervention period will be mixed and assessed at the end of the study. The raters will be blinded to which period the video originates from
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention - Video debriefing (Experimental): Baseline period (year 1): Standard practice. Intervention period (year 2-3): All teams will be assigned to video debriefing.
  Interventions: Behavioral: Video debriefing

INTERVENTIONS:
Behavioral: Video debriefing — Obstetric teams will review their own performance on video in a debriefing session to improve future performance.

SUMMARY:
Postpartum hemorrhage continues to be the leading cause of maternal morbidity and mortality worldwide. Successful management of postpartum hemorrhage requires not only administration of the right medicine, but also a rapid and coordinated response from a multi-professional team. A prerequisite for this is that the individuals are well trained, which the investigators believe can be improved by video debriefing of real-life events.

The purpose of this study is to improve obstetric teams management of postpartum hemorrhage using video recordings of real-life events in post event debriefings.

Cameras are placed in the ceiling of all delivery rooms to record obstetric teams' management of postpartum hemorrhage. Video recording requires informed consent from all participants. After an event, the team will review their own performance on video in a debriefing session to improve future performance.

DETAILED DESCRIPTION:
Background:

Video review was first introduced in healthcare in the 1980s to improve emergency teams' management of critical situations by having them review their own performance on video in a debriefing session. Video debriefing offers an opportunity to review the care delivered in high-stake, high-risk, and time-critical situations. Video debriefing has been found to improve the performance of neonatal resuscitation teams and trauma teams; however, video debriefing has not generally been accepted in the delivery ward. A recent PhD project developed a method for systematically filming obstetric emergencies, in two Danish hospitals, where informed consent had been obtained from all participants. In addition, the project developed a method for systematically assessing obstetric teams' clinical performance during postpartum hemorrhage

The aim of the study is to examine the effect of real-life video debriefing on obstetric teams' management of major postpartum hemorrhage.

Material and methods:

The study will be conducted at two Danish hospitals, Aarhus University Hospital (5,000 deliveries per year) and Horsens Regional Hospital (2,300 deliveries per year).

All delivery rooms have been equipped with an automatic recording system that enables filming of all postpartum hemorrhage. Video recording requires informed consent from all participants. Women expecting to deliver will be invited to provide informed consent for video recording. If a woman declines the invitation, the cameras will be covered up according to our protocol. If video recording occurs, all participants will be asked to give informed consent again.

Video debriefing will be conducted by educated facilitators of debriefing. Debriefings will follow a protocol and will focus on teams' clinical performance and non-technical skills. The main focus of the debriefing protocol will be clinical debriefing with a main goal of improving clinical performance and patient care.

Videos will be included as follows: 1) Baseline video inclusion, before introducing real-life video debriefings of team performance; 2) During the start-up of the debriefings in an exploratory study; 3) After real-life video debriefings have been introduced as standard procedure.

Perspectives:

This project is the first to evaluate the implementation, feasibility and use of real-life video debriefing in obstetric care. Results from this project can revolutionize the ability to learn from clinical cases and can guide how video can be introduced in ways acceptable to women, relatives and healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Women with major postpartum hemorrhage (1.0 liter or more).

Exclusion Criteria:

* Language difficulties requiring an interpreter or translator

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical performance | All videos will be assessed 2.5 years (autumn 2023)
  Videos will be assessed by raters using the TeamOBS-PPH checklist (Brogaard L et al, Development of the TeamOBS-PPH - targeting clinical performance in postpartum hemorrhage, 2018)

SECONDARY OUTCOMES:
Non-technical performance | All videos will be assessed 2.5 years (autumn 2023)
  Videos will be assessed by raters using the AOTP checklist.
Maternal birth characteristics. Time of day. | Data will be assessed 2.5 years (autumn 2023)
  - Day/Night
Maternal birth characteristics. Blood loss. | Data will be assessed 2.5 years (autumn 2023)
  - Total blood loss (ml)
Maternal birth characteristics. GA. | Data will be assessed 2.5 years (autumn 2023)
  - Gestational age
Maternal birth characteristics. Birth length (>18 hours). | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal birth characteristics. Epidural | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal birth characteristics. Oxytocin. | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal birth characteristics. Induction. | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal birth characteristics. Twin pregnancy. | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal characteristics additional. Age. | Data will be assessed 2.5 years (autumn 2023)
  - Years
Maternal characteristics additional. BMI. | Data will be assessed 2.5 years (autumn 2023)
  - BMI
Maternal characteristics additional. Previous postpartum hemorrhage. | Data will be assessed 2.5 years (autumn 2023)
  - Yes/No
Maternal characteristics additional. Previous births | Data will be assessed 2.5 years (autumn 2023)
  - Number
Team characteristics. Team size. | Data will be assessed 2.5 years (autumn 2023)
  - Number of team members involved
Team characteristics. Hospital. | Data will be assessed 2.5 years (autumn 2023)
  - Regional / University
Neonatal characteristics. Mean birth weight. | Data will be assessed 2.5 years (autumn 2023)
  - Grams
Implementation of video debriefing | Data will be assessed 2.5 years (autumn 2023)
  Number of debriefing sessions performed (in total / per participant / failed attempted sessions).

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Horsens Regional Hospital, Horsens

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will be publicly available in an anonymized form using an open data repository.
Time Frame: Study protocol is available at the projects homepage www.teamobs.dk.
  Trial related documents and data will be available when results are published and until three years after publication of the last study results.
Access Criteria: Interested parties will be able to request the data by contacting the trial sponsor.

REFERENCES:
- [Result] Brogaard L, Kierkegaard O, Hvidman L, Jensen KR, Musaeus P, Uldbjerg N, Manser T. The importance of non-technical performance for teams managing postpartum haemorrhage: video review of 99 obstetric teams. BJOG. 2019 Jul;126(8):1015-1023. doi: 10.1111/1471-0528.15655. Epub 2019 Mar 27. PMID 30771263
- [Result] Brogaard L, Hvidman L, Hinshaw K, Kierkegaard O, Manser T, Musaeus P, Arafeh J, Daniels KI, Judy AE, Uldbjerg N. Development of the TeamOBS-PPH - targeting clinical performance in postpartum hemorrhage. Acta Obstet Gynecol Scand. 2018 Jun;97(6):677-687. doi: 10.1111/aogs.13336. Epub 2018 Apr 2. PMID 29485679